CLINICAL TRIAL: NCT04754217
Title: Valved Graft Post-Market Clinical Follow-up Study
Brief Title: Valved Graft PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10386
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Disease; Ascending Aorta Abnormality; Aortic Dissection
Keywords: Aortic Root Replacement; Ascending Aorta Replacement; Valved Graft; CAVGJ; VAVGJ
MeSH Terms: conditions — Aortic Valve Disease; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: VAVGJ
  Interventions: Device: VAVGJ
- Group 2: CAVGJ
  Interventions: Device: CAVGJ

INTERVENTIONS:
Device: VAVGJ — Replacement of the aortic valve and ascending aorta
  Groups: Group 1
Device: CAVGJ — Replacement of the aortic valve and ascending aorta
  Groups: Group 2

SUMMARY:
Multicenter, global, prospective, non-randomized, interventional, post-market trial. All subjects enrolled will receive an Abbott Valved Graft device.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery including the implant of a VAVGJ or CAVGJ for native or prosthetic valve replacement

Exclusion Criteria:

* anticoagulation therapy intolerant
* active endocarditis
* anatomical or medical, surgical, psychological or social contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll male and female subjects who will be undergoing replacement of a native or prosthetic aortic heart valve and ascending aorta.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
annualized event rate of all-cause mortality | 5 Years
  Primary Safety Endpoint
annualized event rate of reintervention | 5 Years
  Primary Effectiveness Endpoint

CONTACTS AND LOCATIONS:
Locations (25):
- United States (5):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - Mission Health & Hospitals, Asheville, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Klinik Floridsdorf, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - CHU de Besancon - Jean Minjoz, Besançon
  - CHRU Lille, Lille
  - Groupe Hospitalier Bichat - Claude Bernard, Paris
- Germany (4):
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Klinikum Links der Weser, Bremen
  - Medizinische Hochschule Hannover, Hanover
- Onassis Cardiac Surgery Center, Athens, Greece
- Italy (3):
  - Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale San Raffaele, Milan
  - Policlinico San Donato, San Donato Milanese
- Poland (4):
  - Wojewodzki Szpital Zespolony w Kielcach, Kielce
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw
- Spain (2):
  - Hospital Universitario del Vinalopó, Elche
  - Hospital Universitario Son Espases, Palma de Mallorca
- James Cook University Hospital, Middlesbrough, United Kingdom